CLINICAL TRIAL: NCT01791868
Title: Randomized and Multicenter Study Assessing the Efficacy of Intravenous Sodium Valproate in Addition to First Line Anti Epileptic Treatment of Generalized Convulsive Status Epilepticus.
Brief Title: Efficacy Study of Intravenous Sodium Valproate in Addition to First Line Anti Epileptic Treatment of Generalized Convulsive Status Epilepticus.
Acronym: VALSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P100148; 2011-006340-75 (EudraCT Number)
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2017-11

CONDITIONS: Generalized Convulsive Status Epilepticus; Intensive Care Unit
Keywords: Generalized convulsive status epilepticus; Sodium valproate; Refractory status epilepticus; Mortality; Epilepsy; Intensive Care Unit; Neurological sequela; Quality of life; Adult
MeSH Terms: conditions — Status Epilepticus; Epilepsy | interventions — Valproic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous sodium valproate (Experimental): Intravenous sodium valproate:
  30 mg/kg during 15 min then 1 mg/kg/h during 12 h
  Interventions: Drug: Intravenous Sodium Valproate
- Intravenous Placebo (Placebo Comparator): Intravenous Placebo:
  NaCl 0,9 % during 15 min at first then during 12 h.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intravenous Sodium Valproate — According to randomization arm, patients will be treated either by intravenous sodium valproate (30 mg/kg during 15 min then 1 mg/kg/h during 12 h) or intravenous placebo. All included patients will benefit from first-line anti epileptic drugs and symptomatic medical care, in agreement with the French Experts Recommendation 2009(RFE 2009).
  Other Names: DEPAKINE®
  Arms: Intravenous sodium valproate
Drug: Placebo — According to randomization arm, patients will be treated either by intravenous sodium valproate (30 mg/kg during 15 min then 1 mg/kg/h during 12 h) or intravenous placebo. All included patients will benefit from first-line anti epileptic drugs and symptomatic medical care, in agreement with the French Experts Recommendation 2009(RFE 2009).
  Other Names: NaCl 0.9%
  Arms: Intravenous Placebo

SUMMARY:
Study Hypothesis Generalized Convulsive Status Epilepticus (GCSE) is a medical emergency associated with an increased morbidity and a prolonged length of hospital stay. Only 50% of patients are discharged from the hospital within the first month after GCSE. Recent Guidelines from Experts highlight the necessity to improve the efficiency of the first line anti-epileptic (AE) therapy.

Intravenous Sodium Valproate (SV) might be an adjuvant AE drug to the recommended first line AEs. Intravenous SV is available, well tolerated and easily injectible but also has pharmacologic properties for reducing the risk of seizures relapses and for being neuroprotective. However, efficacy of intravenous as an adjuvant therapy in GCSE has never been properly assessed.

Primary Purpose The primary purpose is to assess if the association of intravenous Sodium Valproate with the recommended treatment for Generalized Convulsive Status Epilepticus increases to 20 % the number of living patients, discharged from the hospital at day 15.

DETAILED DESCRIPTION:
Patient admitted Intensive Care Unit (ICU) for a Generalized Convulsive Status Epilepticus (GCSE) will be randomized if they fulfil the inclusion criteria and after the written informed consent is obtained from the patient's next of kin. In clack of closed relatives, patients could be included according to the French Health Code for Case of medical emergency. In this situation, patient's consent should be then obtained as soon as possible According to randomization arm, patients will be treated either by intravenous sodium valproate (30 mg/kg during 15 min then 1 mg/kg/h during 12 h) or intravenous placebo. All included patients will benefit from first-line anti epileptic drugs and symptomatic medical care, in agreement with the Experts recommendation (RFE 2009).

From day-1 to day-15, level consciousness(Glasgow Coma Scale, Richmond Agitation Sedation Scale), delirium (Confusion Assessment Method For Intensive Care Unit), reoccurrence of seizure, vital signs, organ dysfunction (Simplified Acute Physiology Score II, Sequential Organ Failure) will be daily assessed.

At day 2, the preventive oral anti-epileptic drug will be prescribed by a neurologist, blinded from randomization.

At Day 15 and Day 30, neurological status, cognitive functions (Mini Mental State Examination, Frontal Assessment Battery, Glasgow Outcome Scale), and quality of life (SF36) will be assessed by a neurologist, also not aware of the randomization.

The number of patients alive and discharged from Hospital day 15 15th day will assessed.

300 patients with GCSE will be randomized, 150 in each arm, in 16 ICUs and over a period of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18.
* Admitted in a participating ICU for generalized convulsive status epilepticus (GCSE) i.e. with persistent or repeated generalized seizures without regaining consciousness over a period of five minutes. provided that the duration of the treatment prior antiepileptic does not exceed:

  * Six hours if GCSE is already controlled at the time of inclusion (= disappearance seizures regardless of the state of consciousness)
  * Twenty-four hours if GCSE persisted or is recurrent.
* Written informed consent collected from close relation or a family member of the patient. Otherwise, inclusion according to French Health Code in case of medical emergency. In this case, the written informed consent of patient has to be collected as soon as possible then. in absence of a close of patient, the patient may be still included. the consent of the prosecution will be collected

Exclusion Criteria:

* Other type of status epilepticus (including atypical form) occured before the onset of anti epileptic.
* Female patient of childbearing age ≥ 18 ans et < 50 ans
* Patient prior treated by depakine in emergency for the GCSE
* The length of stay in hospital expected before the occurrence of GCSE > 15 days.
* Expected Length of stay in ICU <12h .
* Hypoxic-ischemic encephalopathy.
* Pregnant women, eclampsia checked by a systematic pregnancy test.
* Pre-existing chronic or acute hepatitis, or Cirrhosis B or C.
* Family history of acute hepatitis, especially drug-related hepatitis
* Other sodium valproate Contraindications : Hypersensitivity to sodium valproate or derivatives, acute or chronic hepatitis; personal or family history of severe hepatitis, in particular drug; hepatic porphyria, mefloquine or hypericum taking.
* life expectancy expected ≤ 3 months.
* Patients already included in another clinical trial on GCSE.
* Non affiliation to a social health care.
* Patients under tutelage.
* Patient has already been included in this protocol and who completed the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Number of patients in ICU for a GCSE discharged alive from the hospital at Day 15. | 15 days
  Increasing by 20 % the number of patients admitted in ICU for a GCSE who will be discharged alive from the hospital at Day 15.

SECONDARY OUTCOMES:
Frequency of refractory status epilepticus | 3 months
  To determine if intravenous SV as an adjuvant anti-epileptic drug, and irrespectively of the cause of GCSE, decreases as frequency of refractory status epilepticus at 3 months without increase in rate of side effects.
Morbidity related to ICU stay | 3 months
  To determine if intravenous SV as an adjuvant anti-epileptic drug, and irrespectively of the cause of GCSE, decreases as morbidity related to ICU stay at 3 months without increase in rate of side effects.
Cognitive dysfunction | 3 months
  To determine if intravenous SV as an adjuvant anti-epileptic drug, and irrespectively of the cause of GCSE, decreases as cognitive dysfunction at 3 months without increase in rate of side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Hervé OUTIN, MD, Principal Investigator — Service de Réanimation Médico Chirurgicale, Hôpital Poissy Saint-Germain en Laye
Locations (1):
- Hôpital Raymond Poincare, Garche, Haute de Seine, France

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Sharshar T, Porcher R, Asfar P, Grimaldi L, Jabot J, Argaud L, Lebert C, Bollaert PE, Harlay ML, Chillet P, Maury E, Santoli F, Blanc P, Sonneville R, Vu DC, Rohaut B, Mazeraud A, Alvarez JC, Navarro V, Clair B, Outin H; Valse investigators and for the Groupe d'Explorations Neurologiques en Reanimation (GENER). Valproic acid as adjuvant treatment for convulsive status epilepticus: a randomised clinical trial. Crit Care. 2023 Jan 9;27(1):8. doi: 10.1186/s13054-022-04292-7. PMID 36624526
- [Derived] Sharshar T, Ben Hadj Salem O, Porcher R, Grimaldi-Bensouda L, Heming N, Clair B, Azabou E, Mazeraud A, Rohaut B, Outin H. Valproic Acid as an Adjuvant Treatment for Generalized Convulsive Status Epilepticus in Adults Admitted to Intensive Care Units: Protocol for a Double-Blind, Multicenter Randomized Controlled Trial. JMIR Res Protoc. 2021 Feb 24;10(2):e22511. doi: 10.2196/22511. PMID 33625371